CLINICAL TRIAL: NCT02863328
Title: Efficacy and Safety of Oral Semaglutide Versus Empagliflozin in Subjects With Type 2 Diabetes Mellitus
Acronym: PIONEER 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4223; 2015-005209-36 (EudraCT Number); U1111-1176-6006 (Other: World Health Organization (WHO))
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 14 mg oral semaglutide (Experimental)
  Interventions: Drug: semaglutide
- 25 mg empagliflozin (Active Comparator)
  Interventions: Drug: empagliflozin

INTERVENTIONS:
Drug: semaglutide — Oral administration once-daily.
  Arms: 14 mg oral semaglutide
Drug: empagliflozin — Oral administration once-daily.
  Arms: 25 mg empagliflozin

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate Efficacy and Safety of Oral Semaglutide versus Empagliflozin in Subjects with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus at least 90 days prior to day of screening
* HbA1c (glycosylated haemoglobin) of 7.0-10.5 % (53-91 mmol/mol) (both inclusive)
* Stable daily dose of metformin (at least 1500 mg or maximum tolerated dose as documented in the subject medical record) at least 90 days prior to the day of screening

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice).For certain specific countries: Additional specific requirements apply
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Family or personal history of Multiple Endocrine Neoplasia Type 2 or Medullary Thyroid Carcinoma
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Any of the following: myocardial infarction, stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening
* Subjects presently classified as being in New York Heart Association Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Subjects with ALT (alanine aminotransferase) above 2.5 x upper normal limit
* Renal impairment defined as Estimated Glomerular Filtration Rate below 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI)
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening. An exception is short-term insulin treatment for acute illness for a total of below or equal to 14 days
* Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ)
* History of diabetic ketoacidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (89):
- United States (42):
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Oviedo, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Perry, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Argentina (3):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Córdoba
- Brazil (3):
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, São Paulo
- Croatia (5):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Krapinske Toplice
  - Novo Nordisk Investigational Site, Pula
  - Novo Nordisk Investigational Site, Virovitica
  - Novo Nordisk Investigational Site, Zagreb
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (5):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Cegléd
  - Novo Nordisk Investigational Site, Nyíregyhaza
  - Novo Nordisk Investigational Site, Salgótarján
  - Novo Nordisk Investigational Site, Szekszárd
- Italy (5):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Lucca
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Siena
- Poland (6):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Puławy
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
  - Novo Nordisk Investigational Site, Zabrze
- Russia (5):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Tyumen
- Serbia (3):
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Spain (8):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Centelles (Barcelona)
  - Novo Nordisk Investigational Site, L'Hospitalet de Llobregat
  - Novo Nordisk Investigational Site, La Roca Del Vallés
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Vic (Barcelona)
- Thailand (2):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Bangkoknoi, Bangkok

REFERENCES:
- [Result] Rodbard HW, Rosenstock J, Canani LH, Deerochanawong C, Gumprecht J, Lindberg SO, Lingvay I, Sondergaard AL, Treppendahl MB, Montanya E; PIONEER 2 Investigators. Oral Semaglutide Versus Empagliflozin in Patients With Type 2 Diabetes Uncontrolled on Metformin: The PIONEER 2 Trial. Diabetes Care. 2019 Dec;42(12):2272-2281. doi: 10.2337/dc19-0883. Epub 2019 Sep 17. PMID 31530666
- [Result] Eliasson B, Ericsson A, Fridhammar A, Nilsson A, Persson S, Chubb B. Long-Term Cost Effectiveness of Oral Semaglutide Versus Empagliflozin and Sitagliptin for the Treatment of Type 2 Diabetes in the Swedish Setting. Pharmacoecon Open. 2022 May;6(3):343-354. doi: 10.1007/s41669-021-00317-z. Epub 2022 Jan 21. PMID 35064550
- [Result] Aroda VR, Bauer R, Christiansen E, Haluzik M, Kallenbach K, Montanya E, Rosenstock J, Meier JJ. Efficacy and safety of oral semaglutide by subgroups of patient characteristics in the PIONEER phase 3 programme. Diabetes Obes Metab. 2022 Jul;24(7):1338-1350. doi: 10.1111/dom.14710. Epub 2022 May 9. PMID 35373893
- [Derived] Pulleyblank R, Larsen NB. Cost-Effectiveness of Semaglutide vs. Empagliflozin, Canagliflozin, and Sitagliptin for Treatment of Patients with Type 2 Diabetes in Denmark: A Decision-Analytic Modelling Study. Pharmacoecon Open. 2023 Jul;7(4):579-591. doi: 10.1007/s41669-023-00416-z. Epub 2023 May 13. PMID 37178435
- [Derived] Mosenzon O, Capehorn MS, De Remigis A, Rasmussen S, Weimers P, Rosenstock J. Impact of semaglutide on high-sensitivity C-reactive protein: exploratory patient-level analyses of SUSTAIN and PIONEER randomized clinical trials. Cardiovasc Diabetol. 2022 Sep 2;21(1):172. doi: 10.1186/s12933-022-01585-7. PMID 36056351
- [Derived] Lingvay I, Capehorn MS, Catarig AM, Johansen P, Lawson J, Sandberg A, Shaw R, Paine A. Efficacy of Once-Weekly Semaglutide vs Empagliflozin Added to Metformin in Type 2 Diabetes: Patient-Level Meta-analysis. J Clin Endocrinol Metab. 2020 Dec 1;105(12):e4593-604. doi: 10.1210/clinem/dgaa577. PMID 32827435
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 108 sites in 12 countries as follows: Argentina (4), Brazil (3), Croatia (4), Greece (7), Hungary (7), Italy (5), Poland (6), Russian Federation (6), Serbia (5), Spain (8), Thailand (3), United States (46). 1 site each in Croatia and Italy, and 2 sites in the United States screened, but didn't randomise any subjects.
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 14 mg: Participants received once-daily oral semaglutide tablets for 52 weeks. Participants started oral semaglutide at 3 mg and were dose escalated in 4-week increments until the final maintenance dose of 14 mg once-daily was reached (i.e. 3 mg from week 0 to week 4, 7 mg from week 4 to week 8, 14 mg from week 8 to week 52).
- Empagliflozin 25 mg: Participants received once-daily empagliflozin tablets for 52 weeks. Participants started empagliflozin at 10 mg for 8 weeks. Participants were treated with empagliflozin 25 mg if their eGFR was greater than or equal to 60 mL/min/1.73m^2 from week 8 to week 52.
Period: Overall Study
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Started (One participant was duplicate, hence removed from 'started' population.) | 411 | 410
Full Analysis Set (FAS) | 411 | 410
Safety Analysis Set (SAS) | 410 | 409
Completed | 400 | 387
Not Completed | 11 | 23
Not completed — Lost to Follow-up | 4 | 10
Not completed — Withdrawal by Subject | 7 | 12
Not completed — Died | 0 | 1

BASELINE CHARACTERISTICS:
Population: FAS comprised of all randomised participants; however, one subject was randomised twice and thereby only included in FAS once.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 411 | 410 | 821
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 58 (10) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 201 | 406
  Male | 206 | 209 | 415
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 108 | 199
  Not Hispanic or Latino | 320 | 302 | 622
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Race: White | 355 | 353 | 708
    Race: Black or African American | 26 | 33 | 59
    Race: Asian | 28 | 21 | 49
    Race: American Indian or Alaska Native | 0 | 0 | 0
    Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 0
    Race: Other | 2 | 3 | 5
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.1 (0.9) | 8.1 (0.9) | 8.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 26. The endpoint was evaluated based on data from the in-trial observation period which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants, however, one participant was randomised twice and thereby included only once in the FAS. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage-point of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Percentage-point of HbA1c
  In-trial: number analyzed (Participants) | 392 | 395
  In-trial | -1.3 (1.1) | -0.9 (0.9)
  On-treatment without rescue medication: number analyzed (Participants) | 347 | 378
  On-treatment without rescue medication | -1.5 (1.1) | -0.9 (0.9)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an analysis of covariance (ANCOVA) model with treatment and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Non-Inferiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand). A value of 0.4% (the non-inferiority margin) was added to imputed values at week 26 for the oral semaglutide treatment arm only; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from the non-inferiority margin (non-inferiority). The non-inferiority margin was 0.4%; Treatment difference = -0.4, 95% CI 2-sided [-0.6 to -0.3] — Oral semaglutide 14 mg - Empagliflozin 25 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Treatment difference = -0.4, 95% CI 2-sided [-0.6 to -0.3] — Oral semaglutide 14 mg - Empagliflozin 25 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; The analysis was based on a mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment and region as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Non-Inferiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication and any effect after premature trial product discontinuation (hypothetical estimand); p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Treatment difference = -0.5, 95% CI 2-sided [-0.7 to -0.4] — Oral semaglutide 14 mg - Empagliflozin 25 mg
Statistical Analysis 4: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment and region as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Treatment difference = -0.5, 95% CI 2-sided [-0.7 to -0.4] — Oral semaglutide 14 mg - Empagliflozin 25 mg

2. Secondary Outcome: Change in Body Weight (Kg)
Description: Change from baseline (week 0) in body weight was evaluated at week 26. The endpoint was evaluated based on data from the in-trial observation period which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants, however, one participant was randomised twice and thereby included only once in the FAS. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Kilogram (Kg)
  In-trial: number analyzed (Participants) | 393 | 396
  In-trial | -3.9 (4.4) | -3.8 (3.8)
  On-treatment without rescue medication: number analyzed (Participants) | 348 | 378
  On-treatment without rescue medication | -4.3 (4.4) | -3.9 (3.8)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment and region as categorical fixed effects and baseline body weight value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.7593, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Treatment difference = -0.1, 95% CI 2-sided [-0.7 to 0.5] — Oral semaglutide 14 mg - Empagliflozin 25 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment and region as categorical fixed effects and the baseline body weight value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p = 0.1358, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Treatment difference = -0.4, 95% CI 2-sided [-1.0 to 0.1] — Oral semaglutide 14 mg - Empagliflozin 25 mg

3. Secondary Outcome: Change in HbA1c (%)
Description: Change from baseline (week 0) in HbA1c was evaluated at week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 384 | 382
Percentage of HbA1c | -1.3 (1.2) [lower limit 1.2] | -0.9 (1.0) [lower limit 1.0]

4. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) in body weight was evaluated at week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 386 | 383
Kg | -4.0 (5.5) [lower limit 5.5] | -3.7 (4.3) [lower limit 4.3]

5. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline (week 0) in fasting plasma glucose was evaluated at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Millimoles per liter (mmol/L)
  Week 26: number analyzed (Participants) | 388 | 391
  Week 26 | -2.01 (2.56) | -2.08 (2.17)
  Week 52: number analyzed (Participants) | 380 | 378
  Week 52 | -2.04 (2.50) | -2.14 (2.36)

6. Secondary Outcome: Change in SMPG : Mean of the 7-point Profile
Description: Change from baseline (week 0) in mean of the 7-point self-measured plasma glucose (SMPG) (i.e. before and after breakfast, lunch and dinner, and at bedtime) profile was evaluated at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
mmol/L
  Week 26: number analyzed (Participants) | 351 | 351
  Week 26 | -2.3 (2.1) | -1.9 (2.1)
  Week 52: number analyzed (Participants) | 334 | 349
  Week 52 | -2.3 (2.3) | -2.1 (2.3)

7. Secondary Outcome: Change in SMPG : Mean Postprandial Increment Over All Meals
Description: Change from baseline (week 0) in mean postprandial glucose increment was evaluated at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
mmol/L
  Week 26: number analyzed (Participants) | 351 | 354
  Week 26 | -0.5 (1.8) | -0.4 (2.0)
  Week 52: number analyzed (Participants) | 335 | 350
  Week 52 | -0.6 (1.8) | -0.4 (1.9)

8. Secondary Outcome: Change in Fasting C-peptide (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting C-peptide (Nanomoles per liter [nmol/L]) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-peptide
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of C-peptide
  week 26: number analyzed (Participants) | 381 | 387
  week 26 | 1.10 (35.7) | 0.89 (29.4)
  week 52: number analyzed (Participants) | 377 | 381
  week 52 | 1.09 (37.2) | 0.92 (31.6)

9. Secondary Outcome: Change in Fasting Insulin (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting insulin (picomoles per liter [pmol/L]) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of insulin
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of insulin
  Week 26: number analyzed (Participants) | 379 | 386
  Week 26 | 1.06 (50.5) | 0.77 (54.1)
  Week 52: number analyzed (Participants) | 376 | 378
  Week 52 | 1.03 (52.8) | 0.77 (53.7)

10. Secondary Outcome: Change in Fasting Pro-insulin (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting pro-insulin (pmol/L) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of pro-insulin
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of pro-insulin
  Week 26: number analyzed (Participants) | 383 | 388
  Week 26 | 0.72 (74.6) | 0.66 (61.9)
  Week 52: number analyzed (Participants) | 377 | 377
  Week 52 | 0.74 (80.5) | 0.69 (57.8)

11. Secondary Outcome: Change in Fasting Glucagon (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting glucagon (picograms per milliliter [pg/mL]) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of glucagon
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of glucagon
  Week 26: number analyzed (Participants) | 385 | 383
  Week 26 | 0.91 (28.0) | 1.01 (27.5)
  Week 52: number analyzed (Participants) | 377 | 376
  Week 52 | 0.89 (27.8) | 0.95 (27.6)

12. Secondary Outcome: Change in HOMA-IR (Ratio to Baseline)
Description: Change from baseline (week 0) in homeostatic model assessment index of insulin resistance (HOMA-IR) (%) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-IR
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of HOMA-IR
  Week 26: number analyzed (Participants) | 376 | 383
  Week 26 | 0.83 (63.8) | 0.61 (58.7)
  Week 52: number analyzed (Participants) | 374 | 374
  Week 52 | 0.81 (64.9) | 0.60 (60.4)

13. Secondary Outcome: Change in HOMA-B (Ratio to Baseline)
Description: Change from baseline (week 0) in homeostatic model assessment index of beta-cell function (HOMA-B) (%) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-B
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of HOMA-B
  Week 26: number analyzed (Participants) | 376 | 383
  Week 26 | 1.67 (69.5) | 1.16 (65.0)
  Week 52: number analyzed (Participants) | 374 | 374
  Week 52 | 1.66 (72.9) | 1.17 (69.9)

14. Secondary Outcome: Change in C-reactive Protein (Ratio to Baseline)
Description: Change from baseline (week 0) in C-reactive protein (milligrams per liter [mg/L]) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-reactive protein
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of C-reactive protein
  Week 26: number analyzed (Participants) | 388 | 395
  Week 26 | 0.69 (121.5) | 0.98 (115.7)
  Week 52: number analyzed (Participants) | 378 | 381
  Week 52 | 0.68 (129.7) | 0.90 (126.3)

15. Secondary Outcome: Change in Body Weight (%)
Description: Relative change from baseline (week 0) in body weight (kg) was evaluated at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Percentage change
  Week 26: number analyzed (Participants) | 393 | 396
  Week 26 | -4.34 (4.51) | -4.14 (4.12)
  Week 52: number analyzed (Participants) | 386 | 383
  Week 52 | -4.38 (5.76) | -4.09 (4.78)

16. Secondary Outcome: Change in Body Mass Index
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Kilograms per square meter (kg/m^2)
  Week 26: number analyzed (Participants) | 392 | 396
  Week 26 | -1.4 (1.6) | -1.4 (1.4)
  Week 52: number analyzed (Participants) | 385 | 383
  Week 52 | -1.5 (2.0) | -1.4 (1.6)

17. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Centimetre (cm)
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Centimetre (cm)
  Week 26: number analyzed (Participants) | 393 | 393
  Week 26 | -3.9 (5.1) | -2.9 (5.0)
  Week 52: number analyzed (Participants) | 386 | 378
  Week 52 | -3.7 (5.5) | -2.9 (5.8)

18. Secondary Outcome: Change in Fasting Total Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting total cholesterol (mmol/L) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of total cholesterol
  Week 26: number analyzed (Participants) | 387 | 393
  Week 26 | 0.96 (18.1) | 1.02 (15.2)
  Week 52: number analyzed (Participants) | 377 | 381
  Week 52 | 0.97 (18.1) | 1.01 (17.1)

19. Secondary Outcome: Change in Fasting LDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting low density lipoprotein (LDL) cholesterol (mmol/L) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of LDL cholesterol
  Week 26: number analyzed (Participants) | 386 | 393
  Week 26 | 0.96 (38.3) | 1.03 (24.6)
  Week 52: number analyzed (Participants) | 377 | 381
  Week 52 | 0.97 (30.1) | 1.03 (27.2)

20. Secondary Outcome: Change in Fasting HDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting high density lipoprotein (HDL) cholesterol (mmol/L) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of HDL cholesterol
  Week 26: number analyzed (Participants) | 387 | 393
  Week 26 | 1.01 (13.0) | 1.07 (15.9)
  Week 52: number analyzed (Participants) | 377 | 381
  Week 52 | 1.01 (13.9) | 1.06 (14.0)

21. Secondary Outcome: Change in Fasting VLDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting very low density lipoprotein (VLDL) cholesterol (mmol/L) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of VLDL cholesterol
  Week 26: number analyzed (Participants) | 387 | 393
  Week 26 | 0.89 (39.0) | 0.91 (34.7)
  Week 52: number analyzed (Participants) | 377 | 381
  Week 52 | 0.89 (39.3) | 0.90 (37.6)

22. Secondary Outcome: Change in Fasting Free Fatty Acids (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting free fatty acids (FFA) (mmol/L) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. Because of an issue with the handling of the blood samples for FFA, all FFA data are considered invalid for this trial; thus, no conclusion with regards to FFA levels can be made based on the FFA data. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FFA
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of FFA
  Week 26: number analyzed (Participants) | 385 | 390
  Week 26 | 0.95 (51.3) | 1.05 (46.9)
  Week 52: number analyzed (Participants) | 380 | 376
  Week 52 | 0.88 (53.0) | 0.97 (49.2)

23. Secondary Outcome: Change in Fasting Triglycerides (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting triglycerides (mmol/L) at week 26 and week 52 is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Ratio of triglycerides
  Week 26: number analyzed (Participants) | 387 | 393
  Week 26 | 0.88 (40.5) | 0.90 (36.1)
  Week 52: number analyzed (Participants) | 377 | 381
  Week 52 | 0.89 (42.3) | 0.90 (39.3)

24. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) ADA Target (Yes/no)
Description: Participants who achieved HbA1c <7.0% (53 mmol/mol) (American Diabetes Association (ADA) target) at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26 and week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  Week 26: number analyzed (Participants) | 392 | 395
  Week 26: Yes | 262 | 158
  Week 26: No | 130 | 237
  Week 52: number analyzed (Participants) | 384 | 382
  Week 52: Yes | 254 | 165
  Week 52: No | 130 | 217

25. Secondary Outcome: Participants Who Achieve HbA1c ≤6.5% (48 mmol/Mol), AACE Target (Yes/no)
Description: Participants who achieved HbA1c ≤6.5% (48 mmol/mol) (American Association of Clinical Endocrinologists (AACE) target) at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26 and week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  Week 26: number analyzed (Participants) | 392 | 395
  Week 26: Yes | 186 | 68
  Week 26: No | 206 | 327
  Week 52: number analyzed (Participants) | 384 | 382
  Week 52: Yes | 182 | 83
  Week 52: No | 202 | 299

26. Secondary Outcome: Participants Who Achieve Weight Loss ≥5% (Yes/no)
Description: Participants who achieved weight loss of ≥5% at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26 and week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  Week 26: number analyzed (Participants) | 393 | 396
  Week 26: Yes | 162 | 143
  Week 26: No | 231 | 253
  Week 52: number analyzed (Participants) | 386 | 383
  Week 52: Yes | 156 | 150
  Week 52: No | 230 | 233

27. Secondary Outcome: Participants Who Achieve Weight Loss ≥10% (Yes/no)
Description: Participants who achieved weight loss of ≥10% at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26 and week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  Week 26: number analyzed (Participants) | 393 | 396
  Week 26: Yes | 49 | 27
  Week 26: No | 344 | 369
  Week 52: number analyzed (Participants) | 386 | 383
  Week 52: Yes | 58 | 30
  Week 52: No | 328 | 353

28. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)
Description: Participants who achieved HbA1c <7.0% (53 mmol/mol) without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain at week 26 and week 52. Severe or BG-confirmed symptomatic hypoglycaemia: an episode, that is severe according to the ADA classification or BG-confirmed by a plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26 and week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  Week 26: number analyzed (Participants) | 392 | 395
  Week 26: Yes | 237 | 141
  Week 26: No | 155 | 254
  Week 52: number analyzed (Participants) | 384 | 382
  Week 52: Yes | 214 | 149
  Week 52: No | 170 | 233

29. Secondary Outcome: Participants Who Achieve HbA1c Reduction ≥1% (10.9 mmol/Mol) and Weight Loss ≥3% (Yes/no)
Description: Participants who achieved HbA1c reduction ≥1%-point and weight loss of ≥3% at week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26 and week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  week 26: number analyzed (Participants) | 392 | 395
  week 26: Yes | 177 | 111
  week 26: No | 215 | 284
  week 52: number analyzed (Participants) | 384 | 382
  week 52: Yes | 164 | 101
  week 52: No | 220 | 281

30. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Additional anti-diabetic medication: use of new anti-diabetic medication for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment (week 26/week 52), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants, however, one participant was randomised twice and thereby included only once in the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  Week 0-26 | 17 | 13
  Week 0-52 | 52 | 56
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment and region as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.3552, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.60 to 1.20] — Oral semaglutide 14 mg / Empagliflozin 25 mg

31. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Rescue medication: use of new antidiabetic medication as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 0) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period. On-treatment without rescue medication observation period: the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Weeks 0-52
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Participants
  Week 0-26 | 8 | 5
  Week 0-52 | 31 | 44
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Empagliflozin 25 mg; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.2250, Cox proportional hazards model — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.47 to 1.19] — Oral semaglutide 14 mg / Empagliflozin 25 mg

32. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAE)
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) with onset in the on-treatment observation period (the time period where participants are considered treated with trial product) and was assessed up to approximately 57 weeks (52-week treatment period plus the 5-week follow-up period).
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Events | 1022 | 948

33. Secondary Outcome: Change in Amylase (Ratio to Baseline)
Description: Change from baseline (week 0) in amylase (units per liter [U/L]) at week 26 and week 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Ratio of amylase
  Week 26: number analyzed (Participants) | 352 | 382
  Week 26 | 1.15 (30.1) | 1.10 (24.8)
  Week 52: number analyzed (Participants) | 330 | 359
  Week 52 | 1.13 (31.5) | 1.11 (26.8)

34. Secondary Outcome: Change in Lipase (Ratio to Baseline)
Description: Change from baseline (week 0) in lipase (U/L) at week 26 and week 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Ratio of lipase
  Week 26: number analyzed (Participants) | 352 | 382
  Week 26 | 1.37 (62.0) | 1.10 (50.8)
  Week 52: number analyzed (Participants) | 330 | 359
  Week 52 | 1.27 (63.6) | 1.07 (47.2)

35. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at week 26 and week 52. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Beats/minute
  Week 26: number analyzed (Participants) | 356 | 383
  Week 26 | 1 (10) | -2 (9)
  Week 52: number analyzed (Participants) | 336 | 364
  Week 52 | 1 (10) | -2 (9)

36. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated at week 26 and week 52. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Millimeters of mercury (mmHg)
  SBP, week 26: number analyzed (Participants) | 357 | 383
  SBP, week 26 | -5 (15) | -5 (14)
  SBP, week 52: number analyzed (Participants) | 337 | 364
  SBP, week 52 | -5 (13) | -4 (15)
  DBP, week 26: number analyzed (Participants) | 357 | 383
  DBP, week 26 | -2 (9) | -3 (9)
  DBP, week 52: number analyzed (Participants) | 337 | 364
  DBP, week 52 | -3 (10) | -3 (9)

37. Secondary Outcome: Change in ECG
Description: Change from baseline (week 0) in electrocardiogram (ECG) was evaluated at week 26 and week 52. Change from baseline results are presented as shift in findings (normal, abnormal and not clinically significant (NCS), and abnormal and clinically significant (CS)) from week 0 to week 26 and week 52. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 238 | 242
  Normal (week 0) to normal (week 26) | 207 | 203
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 238 | 242
  Normal (week 0) to abnormal NCS (week 26) | 30 | 37
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 238 | 242
  Normal (week 0) to abnormal CS (week 26) | 1 | 2
  Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 147 | 151
  Abnormal NCS (week 0) to normal (week 26) | 50 | 41
  Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 147 | 151
  Abnormal NCS (week 0) to abnormal NCS (week 26) | 97 | 110
  Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 147 | 151
  Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0
  Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 4 | 1
  Abnormal CS (week 0) to normal (week 26) | 1 | 0
  Abnormal CS (week 0) CS to abnormal NCS (week 26): number analyzed (Participants) | 4 | 1
  Abnormal CS (week 0) CS to abnormal NCS (week 26) | 2 | 0
  Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 4 | 1
  Abnormal CS (week 0) to abnormal CS (week 26) | 1 | 1
  Normal (week 0) to normal (week 52): number analyzed (Participants) | 235 | 235
  Normal (week 0) to normal (week 52) | 196 | 194
  Normal (week 0) to abnormal NCS (week 52): number analyzed (Participants) | 235 | 235
  Normal (week 0) to abnormal NCS (week 52) | 39 | 39
  Normal (week 0) to abnormal CS (week 52): number analyzed (Participants) | 235 | 235
  Normal (week 0) to abnormal CS (week 52) | 0 | 2
  Abnormal (week 0) NCS to normal (week 52): number analyzed (Participants) | 145 | 144
  Abnormal (week 0) NCS to normal (week 52) | 46 | 45
  Abnormal (week 0) NCS to abnormal NCS (week 52): number analyzed (Participants) | 145 | 144
  Abnormal (week 0) NCS to abnormal NCS (week 52) | 98 | 97
  Abnormal (week 0) NCS to abnormal CS (week 52): number analyzed (Participants) | 145 | 144
  Abnormal (week 0) NCS to abnormal CS (week 52) | 1 | 2
  Abnormal CS (week 0) to normal (week 52): number analyzed (Participants) | 4 | 1
  Abnormal CS (week 0) to normal (week 52) | 1 | 0
  Abnormal CS (week 0) to abnormal NCS (week 52): number analyzed (Participants) | 4 | 1
  Abnormal CS (week 0) to abnormal NCS (week 52) | 2 | 0
  Abnormal CS (week 0) to abnormal CS (week 52): number analyzed (Participants) | 4 | 1
  Abnormal CS (week 0) to abnormal CS (week 52) | 1 | 1

38. Secondary Outcome: Change in Physical Examination
Description: The physical examination findings (normal, abnormal NCS and abnormal CS) of the participants at week -2 and week 52 are presented for the following examinations: Cardiovascular system, Nervous system (central and peripheral); Gastrointestinal system, incl. mouth; General appearance; Head (ears, eyes, nose), throat, neck; Lymph node palpation; Musculoskeletal system; Respiratory system; Skin; Thyroid gland. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week -2, week 52
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Participants
  Cardiovascular system (week -2): Normal | 381 | 372
  Cardiovascular system (week -2): Abnormal NCS | 24 | 34
  Cardiovascular system (week -2): Abnormal CS | 5 | 3
  Cardiovascular system (week 52): number analyzed (Participants) | 385 | 382
  Cardiovascular system (week 52): Normal | 360 | 351
  Cardiovascular system (week 52): Abnormal NCS | 21 | 29
  Cardiovascular system (week 52): Abnormal CS | 4 | 2
  Nervous system (week -2): Normal | 390 | 376
  Nervous system (week -2): Abnormal NCS | 20 | 30
  Nervous system (week -2): Abnormal CS | 0 | 3
  Nervous system (week 52): number analyzed (Participants) | 385 | 383
  Nervous system (week 52): Normal | 371 | 365
  Nervous system (week 52): Abnormal NCS | 13 | 17
  Nervous system (week 52): Abnormal CS | 1 | 1
  Gastrointestinal system (week -2): Normal | 387 | 384
  Gastrointestinal system (week -2): Abnormal NCS | 23 | 24
  Gastrointestinal system (week -2): Abnormal CS | 0 | 1
  Gastrointestinal system (week 52): number analyzed (Participants) | 385 | 382
  Gastrointestinal system (week 52): Normal | 366 | 360
  Gastrointestinal system (week 52): Abnormal NCS | 18 | 22
  Gastrointestinal system (week 52): Abnormal CS | 1 | 0
  General appearance (week -2): Normal | 354 | 354
  General appearance (week -2): Abnormal NCS | 47 | 49
  General appearance (week -2): Abnormal CS | 9 | 6
  General appearance (week 52): number analyzed (Participants) | 385 | 383
  General appearance (week 52): Normal | 345 | 338
  General appearance (week 52): Abnormal NCS | 36 | 41
  General appearance (week 52): Abnormal CS | 4 | 4
  Head, throat, neck (week -2): Normal | 389 | 382
  Head, throat, neck (week -2): Abnormal NCS | 18 | 26
  Head, throat, neck (week -2): Abnormal CS | 3 | 1
  Head, throat, neck (week 52): number analyzed (Participants) | 385 | 383
  Head, throat, neck (week 52): Normal | 376 | 362
  Head, throat, neck (week 52): Abnormal NCS | 8 | 19
  Head, throat, neck (week 52): Abnormal CS | 1 | 2
  Lymph node palpation (week -2): Normal | 409 | 409
  Lymph node palpation (week -2): Abnormal NCS | 1 | 0
  Lymph node palpation (week -2): Abnormal CS | 0 | 0
  Lymph node palpation (week 52): number analyzed (Participants) | 385 | 381
  Lymph node palpation (week 52): Normal | 385 | 381
  Lymph node palpation (week 52): Abnormal NCS | 0 | 0
  Lymph node palpation (week 52): Abnormal CS | 0 | 0
  Musculoskeletal system (week -2): Normal | 389 | 384
  Musculoskeletal system (week -2): Abnormal NCS | 18 | 25
  Musculoskeletal system (week -2): Abnormal CS | 3 | 0
  Musculoskeletal system (week 52): number analyzed (Participants) | 385 | 383
  Musculoskeletal system (week 52): Normal | 370 | 363
  Musculoskeletal system (week 52): Abnormal NCS | 15 | 20
  Musculoskeletal system (week 52): Abnormal CS | 0 | 0
  Respiratory system (week -2): Normal | 400 | 403
  Respiratory system (week -2): Abnormal NCS | 9 | 6
  Respiratory system (week -2): Abnormal CS | 1 | 0
  Respiratory system (week 52): number analyzed (Participants) | 385 | 382
  Respiratory system (week 52): Normal | 375 | 378
  Respiratory system (week 52): Abnormal NCS | 8 | 4
  Respiratory system (week 52): Abnormal CS | 2 | 0
  Skin (week -2): Normal | 357 | 354
  Skin (week -2): Abnormal NCS | 50 | 53
  Skin (week -2): Abnormal CS | 3 | 2
  Skin (week 52): number analyzed (Participants) | 385 | 383
  Skin (week 52): Normal | 346 | 340
  Skin (week 52): Abnormal NCS | 37 | 42
  Skin (week 52): Abnormal CS | 2 | 1
  Thyroid gland (week -2): Normal | 399 | 389
  Thyroid gland (week -2): Abnormal NCS | 11 | 18
  Thyroid gland (week -2): Abnormal CS | 0 | 2
  Thyroid gland (week 52): number analyzed (Participants) | 385 | 383
  Thyroid gland (week 52): Normal | 376 | 367
  Thyroid gland (week 52): Abnormal NCS | 9 | 16
  Thyroid gland (week 52): Abnormal CS | 0 | 0

39. Secondary Outcome: Change in Eye Examination
Description: The eye examination findings (normal, abnormal NCS and abnormal CS) of the participants at baseline (week -2) and week 52 are presented. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week -2, week 52
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Participants
  Left eye (week -2): number analyzed (Participants) | 409 | 407
  Left eye (week -2): Normal | 295 | 295
  Left eye (week -2): Abnormal NCS | 107 | 102
  Left eye (week -2): Abnormal CS | 7 | 10
  Left eye (week 52): number analyzed (Participants) | 375 | 372
  Left eye (week 52): Normal | 264 | 269
  Left eye (week 52): Abnormal NCS | 103 | 93
  Left eye (week 52): Abnormal CS | 8 | 10
  Right eye (week -2): number analyzed (Participants) | 409 | 409
  Right eye (week -2): Normal | 294 | 293
  Right eye (week -2): Abnormal NCS | 109 | 107
  Right eye (week -2): Abnormal CS | 6 | 9
  Right eye (week 52): number analyzed (Participants) | 374 | 373
  Right eye (week 52): Normal | 267 | 269
  Right eye (week 52): Abnormal NCS | 96 | 93
  Right eye (week 52): Abnormal CS | 11 | 11

40. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide binding antibodies anytime during post-baseline visits (week 0 to week 57) are presented. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 403
Participants | 2

41. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide neutralising antibodies anytime during post-baseline visits (week 0 to week 57) are presented. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 403
Participants | 0

42. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide binding antibodies cross reacting with native glucagon-like peptide-1 (GLP-1) anytime during post-baseline visits (week 0 to week 57) are presented. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 403
Participants | 0

43. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide neutralising antibodies cross reacting with native GLP-1 anytime during post-baseline visits (week 0 to week 57) are presented. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 403
Participants | 0

44. Secondary Outcome: Anti-semaglutide Binding Antibody Levels
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. It is based on the data from participants who were measured with anti-semaglutide antibodies anytime during post-baseline visits (week 0 to week 57). Results are presented as percentage of bound radioactivity-labelled semaglutide /total added radioactivity-labelled semaglutide (%B/T). The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: Overall number of participants analysed = participants who were found positive for anti-semaglutide antibodies.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 2
%B/T
  Week 4: number analyzed (Participants) | 1
  Week 4 | 2.75 (0.00)
  Week 8: number analyzed (Participants) | 1
  Week 8 | 2.17 (0.00)
  Week 14: number analyzed (Participants) | 0
  Week 26: number analyzed (Participants) | 0
  Week 38: number analyzed (Participants) | 0
  Week 52: number analyzed (Participants) | 0
  Week 57: number analyzed (Participants) | 0

45. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment-emergent hypoglycaemia is an episode with onset in the on-treatment observation period (the time period where participants are considered treated with trial product) and was assessed up to approximately 57 weeks (52-week treatment period plus the 5-week follow-up period). Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Episodes | 10 | 9

46. Secondary Outcome: Participants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes (Yes/no)
Description: Number of participants with treatment-emergent severe or BG-confirmed symptomatic hypoglycaemic episodes was recorded during week 0-57. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-57
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 410 | 409
Participants | 7 | 8

47. Secondary Outcome: Semaglutide Plasma Concentrations for Population PK Analyses
Description: Semaglutide plasma concentrations were measured after 25 minutes post-dose at week 4, 26 and 52. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 411
Nanomoles per liter (nmol/L)
  Week 4: number analyzed (Participants) | 392
  Week 4 | 3.5 (84.5)
  Week 26: number analyzed (Participants) | 348
  Week 26 | 15.6 (112.4)
  Week 52: number analyzed (Participants) | 331
  Week 52 | 14.4 (136.6)

48. Secondary Outcome: SNAC Plasma Concentrations
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Sodium N-[8-(2-hydroxybenzoyl) amino]caprylate (SNAC) plasma concentrations were measured after 25 and 40 minutes post-dose at week 4, 26 and 52. Results are based on the data from the on-treatment observation period. On-treatment observation period: the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 411
Nanograms per milliliter (ng/mL)
  Week 4: 25 minutes post-dose: number analyzed (Participants) | 390
  Week 4: 25 minutes post-dose | 559 (224.6)
  Week 4: 40 minutes post-dose: number analyzed (Participants) | 392
  Week 4: 40 minutes post-dose | 375 (210.4)
  Week 26: 25 minutes post-dose: number analyzed (Participants) | 350
  Week 26: 25 minutes post-dose | 474 (272.7)
  Week 26: 40 minutes post-dose: number analyzed (Participants) | 349
  Week 26: 40 minutes post-dose | 373 (200.6)
  Week 52: 25 minutes post-dose: number analyzed (Participants) | 331
  Week 52: 25 minutes post-dose | 448 (377.5)
  Week 52: 40 minutes post-dose: number analyzed (Participants) | 331
  Week 52: 40 minutes post-dose | 301 (290.2)

49. Secondary Outcome: Change in Short Form Health Survey Version 2.0 (SF-36v2™, Acute Version) Health Survey: Scores From the 8 Domains and Summaries of the Physical Component Score (PCS) and the Mental Component Score (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at weeks 26 and 52. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Score on a scale
  Week 26: Physical Functioning: number analyzed (Participants) | 392 | 396
  Week 26: Physical Functioning | 0.87 (7.35) | 0.99 (7.11)
  Week 52: Physical Functioning: number analyzed (Participants) | 386 | 383
  Week 52: Physical Functioning | 0.57 (6.79) | 0.84 (7.32)
  Week 26: Role functioning: number analyzed (Participants) | 392 | 396
  Week 26: Role functioning | 0.07 (6.82) | 0.56 (8.36)
  Week 52: Role functioning: number analyzed (Participants) | 386 | 382
  Week 52: Role functioning | -0.61 (6.78) | 0.52 (7.93)
  Week 26: Bodily pain: number analyzed (Participants) | 392 | 396
  Week 26: Bodily pain | -0.32 (9.77) | 1.04 (9.53)
  Week 52: Bodily pain: number analyzed (Participants) | 386 | 383
  Week 52: Bodily pain | -0.33 (10.07) | 1.20 (9.54)
  Week 26: General health: number analyzed (Participants) | 392 | 396
  Week 26: General health | 2.26 (6.59) | 1.36 (6.56)
  Week 52: General health: number analyzed (Participants) | 386 | 383
  Week 52: General health | 2.47 (7.35) | 1.86 (7.66)
  Week 26: Vitality: number analyzed (Participants) | 392 | 396
  Week 26: Vitality | 0.66 (7.58) | 0.49 (7.60)
  Week 52: Vitality: number analyzed (Participants) | 386 | 383
  Week 52: Vitality | 0.83 (7.72) | 1.15 (7.48)
  Week 26: Social functioning: number analyzed (Participants) | 392 | 396
  Week 26: Social functioning | 0.50 (7.28) | -0.54 (8.15)
  Week 52: Social functioning: number analyzed (Participants) | 386 | 383
  Week 52: Social functioning | -0.18 (8.35) | -0.54 (8.63)
  Week 26: Role emotional: number analyzed (Participants) | 392 | 396
  Week 26: Role emotional | 0.67 (9.47) | 0.53 (9.49)
  Week 52: Role emotional: number analyzed (Participants) | 386 | 382
  Week 52: Role emotional | 0.30 (9.63) | 0.42 (9.93)
  Week 26: Mental health: number analyzed (Participants) | 392 | 396
  Week 26: Mental health | 0.94 (8.06) | -0.03 (8.70)
  Week 52: Mental health: number analyzed (Participants) | 386 | 383
  Week 52: Mental health | 0.29 (8.71) | -0.03 (9.21)
  Week 26: PCS: number analyzed (Participants) | 392 | 396
  Week 26: PCS | 0.53 (6.36) | 1.21 (6.39)
  Week 52: PCS: number analyzed (Participants) | 386 | 382
  Week 52: PCS | 0.44 (6.26) | 1.36 (6.50)
  Week 26: MCS: number analyzed (Participants) | 392 | 396
  Week 26: MCS | 0.83 (7.54) | -0.23 (8.40)
  Week 52: MCS: number analyzed (Participants) | 386 | 382
  Week 52: MCS | 0.35 (8.36) | -0.09 (8.64)

50. Secondary Outcome: Change in CoEQ: Scores From the 4 Domains and the 19 Items
Description: Change from baseline (week 0) in Control of Eating Questionnaire (CoEQ) was evaluated at weeks 26 and 52. The CoEQ comprised 19 items to assess the intensity and type of food cravings, as well as subjective sensation of appetite and mood, with the 4 domains: 'craving control' (items 9-12, 19), 'positive mood' (items 5-8), 'craving for savoury' (items 4, 16-18) and 'craving for sweet' (items 3, 13-15). The 19 items were scored on an 11-point graded response scale ranging from 10 to 0, with items relating to each of the 4 domains being averaged to create a final score. A low score in the domains 'craving for sweet and 'craving for savoury' represents a low level of craving; whereas a high score in the domains 'craving control' and 'positive mood' represents good control and a good mood, respectively. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 411 | 410
Score on a scale
  Week 26: Craving control: number analyzed (Participants) | 392 | 396
  Week 26: Craving control | 0.46 (2.60) | 0.21 (2.26)
  Week 52: Craving control: number analyzed (Participants) | 386 | 383
  Week 52: Craving control | 0.44 (2.54) | 0.18 (2.38)
  Week 26: Positive Mood: number analyzed (Participants) | 392 | 396
  Week 26: Positive Mood | 0.08 (1.52) | 0.19 (1.62)
  Week 52: Positive Mood: number analyzed (Participants) | 386 | 383
  Week 52: Positive Mood | 0.15 (1.75) | 0.17 (1.64)
  Week 26: Craving for Savoury: number analyzed (Participants) | 392 | 395
  Week 26: Craving for Savoury | -0.68 (2.13) | -0.54 (2.05)
  Week 52: Craving for Savoury: number analyzed (Participants) | 386 | 383
  Week 52: Craving for Savoury | -0.66 (2.16) | -0.44 (2.14)
  Week 26: Craving for Sweet: number analyzed (Participants) | 392 | 395
  Week 26: Craving for Sweet | -0.25 (2.15) | -0.21 (2.04)
  Week 52: Craving for Sweet: number analyzed (Participants) | 386 | 383
  Week 52: Craving for Sweet | -0.21 (2.23) | -0.17 (2.13)
  Week 26: 1.Feeling of hunger: number analyzed (Participants) | 392 | 396
  Week 26: 1.Feeling of hunger | -0.80 (2.69) | -0.09 (2.59)
  Week 52: 1.Feeling of hunger: number analyzed (Participants) | 386 | 383
  Week 52: 1.Feeling of hunger | -0.60 (2.82) | 0.07 (2.56)
  Week 26: 2.Feeling of fullness: number analyzed (Participants) | 392 | 395
  Week 26: 2.Feeling of fullness | 0.40 (2.65) | 0.29 (2.63)
  Week 52: 2.Feeling of fullness: number analyzed (Participants) | 386 | 383
  Week 52: 2.Feeling of fullness | 0.35 (2.75) | 0.06 (2.67)
  Week 26: 3.Desire to eat sweet foods: number analyzed (Participants) | 392 | 396
  Week 26: 3.Desire to eat sweet foods | -0.35 (3.04) | -0.22 (2.95)
  Week 52: 3.Desire to eat sweet foods: number analyzed (Participants) | 386 | 383
  Week 52: 3.Desire to eat sweet foods | -0.36 (3.23) | -0.18 (2.85)
  Week 26: 4.Desire to eat savoury foods: number analyzed (Participants) | 392 | 396
  Week 26: 4.Desire to eat savoury foods | -0.82 (2.99) | -0.56 (3.09)
  Week 52: 4.Desire to eat savoury foods: number analyzed (Participants) | 386 | 383
  Week 52: 4.Desire to eat savoury foods | -0.82 (3.15) | -0.57 (2.93)
  Week 26: 5.Feeling of happiness: number analyzed (Participants) | 392 | 396
  Week 26: 5.Feeling of happiness | 0.00 (2.24) | 0.21 (2.31)
  Week 52: 5.Feeling of happiness: number analyzed (Participants) | 386 | 383
  Week 52: 5.Feeling of happiness | 0.13 (2.61) | 0.21 (2.36)
  Week 26: 6.Feeling of anxiousness: number analyzed (Participants) | 392 | 396
  Week 26: 6.Feeling of anxiousness | -0.21 (2.92) | -0.31 (3.22)
  Week 52: 6.Feeling of anxiousness: number analyzed (Participants) | 386 | 383
  Week 52: 6.Feeling of anxiousness | -0.19 (3.03) | -0.21 (3.02)
  Week 26: 7.Feeling of alertness: number analyzed (Participants) | 392 | 396
  Week 26: 7.Feeling of alertness | 0.01 (2.68) | 0.02 (2.57)
  Week 52: 7.Feeling of alertness: number analyzed (Participants) | 385 | 383
  Week 52: 7.Feeling of alertness | 0.07 (2.73) | 0.08 (2.63)
  Week 26: 8.Feeling of contentment: number analyzed (Participants) | 392 | 395
  Week 26: 8.Feeling of contentment | 0.08 (2.37) | 0.22 (2.42)
  Week 52: 8.Feeling of contentment: number analyzed (Participants) | 386 | 383
  Week 52: 8.Feeling of contentment | 0.23 (2.54) | 0.17 (2.30)
  Week 26: 9.Food cravings during 7 days: number analyzed (Participants) | 392 | 396
  Week 26: 9.Food cravings during 7 days | -0.43 (3.25) | -0.03 (3.03)
  Week 52: 9.Food cravings during 7 days: number analyzed (Participants) | 386 | 383
  Week 52: 9.Food cravings during 7 days | -0.42 (3.23) | -0.17 (2.98)
  Week 26: 10.Strength of food cravings: number analyzed (Participants) | 392 | 396
  Week 26: 10.Strength of food cravings | -0.27 (3.11) | -0.18 (2.97)
  Week 52: 10.Strength of food cravings: number analyzed (Participants) | 386 | 383
  Week 52: 10.Strength of food cravings | -0.32 (3.13) | -0.14 (3.01)
  Week 26: 11.Difficulty to resist food cravings: number analyzed (Participants) | 392 | 396
  Week 26: 11.Difficulty to resist food cravings | -0.47 (3.41) | -0.35 (3.18)
  Week 52: 11.Difficulty to resist food cravings: number analyzed (Participants) | 386 | 383
  Week 52: 11.Difficulty to resist food cravings | -0.33 (3.26) | -0.30 (3.24)
  Week 26: 12.Eating in response to food cravings: number analyzed (Participants) | 391 | 396
  Week 26: 12.Eating in response to food cravings | -0.19 (2.94) | -0.12 (2.75)
  Week 52: 12.Eating in response to food cravings: number analyzed (Participants) | 385 | 383
  Week 52: 12.Eating in response to food cravings | -0.17 (2.97) | -0.01 (2.93)
  Week 26: 13.Cravings for chocolate: number analyzed (Participants) | 392 | 395
  Week 26: 13.Cravings for chocolate | -0.10 (3.03) | -0.26 (3.02)
  Week 52: 13.Cravings for chocolate: number analyzed (Participants) | 386 | 383
  Week 52: 13.Cravings for chocolate | 0.08 (3.13) | -0.12 (3.00)
  Week 26: 14.Cravings for other sweet foods: number analyzed (Participants) | 392 | 395
  Week 26: 14.Cravings for other sweet foods | -0.39 (2.91) | -0.36 (2.94)
  Week 52: 14.Cravings for other sweet foods: number analyzed (Participants) | 386 | 383
  Week 52: 14.Cravings for other sweet foods | -0.33 (2.90) | -0.24 (3.13)
  Week 26: 15.Cravings for fruit or fruit juice: number analyzed (Participants) | 392 | 395
  Week 26: 15.Cravings for fruit or fruit juice | -0.15 (3.29) | 0.01 (3.11)
  Week 52: 15.Cravings for fruit or fruit juice: number analyzed (Participants) | 386 | 383
  Week 52: 15.Cravings for fruit or fruit juice | -0.22 (3.31) | -0.15 (3.14)
  Week 26: 16.Cravings for dairy foods: number analyzed (Participants) | 392 | 395
  Week 26: 16.Cravings for dairy foods | -0.48 (3.05) | -0.43 (2.88)
  Week 52: 16.Cravings for dairy foods: number analyzed (Participants) | 386 | 383
  Week 52: 16.Cravings for dairy foods | -0.42 (3.11) | -0.16 (2.92)
  Week 26: 17.Cravings for starchy foods: number analyzed (Participants) | 392 | 395
  Week 26: 17.Cravings for starchy foods | -0.81 (2.99) | -0.59 (2.64)
  Week 52: 17.Cravings for starchy foods: number analyzed (Participants) | 386 | 383
  Week 52: 17.Cravings for starchy foods | -0.78 (3.04) | -0.51 (2.99)
  Week 26: 18.Cravings for savoury foods: number analyzed (Participants) | 392 | 395
  Week 26: 18.Cravings for savoury foods | -0.61 (3.02) | -0.56 (2.93)
  Week 52: 18.Cravings for savoury foods: number analyzed (Participants) | 386 | 383
  Week 52: 18.Cravings for savoury foods | -0.60 (2.92) | -0.50 (3.09)
  Week 26: 19.Difficulty to control eating general: number analyzed (Participants) | 391 | 395
  Week 26: 19.Difficulty to control eating general | -0.90 (3.09) | -0.36 (2.79)
  Week 52: 19.Difficulty to control eating general: number analyzed (Participants) | 385 | 383
  Week 52: 19.Difficulty to control eating general | -0.97 (3.01) | -0.27 (2.82)

ADVERSE EVENTS:
Time Frame: Week 0 to week 57 (52 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 14 mg | Empagliflozin 25 mg
All-Cause Mortality (participants affected / at risk) | 0/410 | 1/409
Serious Adverse Events (participants affected / at risk) | 27/410 | 37/409
Other Adverse Events (participants affected / at risk) | 128/410 | 44/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=410) | Empagliflozin 25 mg (N=409)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
CANVAS syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Head deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypocoagulable state (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=410) | Empagliflozin 25 mg (N=409)
Decreased appetite (Metabolism and nutrition disorders) | 21 (21) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 38 (48) | 13 (17)
Influenza (Infections and infestations) | 8 (8) | 21 (23)
Nausea (Gastrointestinal disorders) | 81 (106) | 10 (12)
Vomiting (Gastrointestinal disorders) | 30 (40) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT02863328/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT02863328/SAP_001.pdf